CLINICAL TRIAL: NCT00467103
Title: Neural Networks and Language Recovery in Aphasia From Stroke: fMRI Studies
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Boston University (Other)
Responsible Party: Sponsor
Other Study IDs: MHBB-006-06S
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Aphasia; Nonfluent Aphasia; Stroke
Keywords: Adult Aphasia; Diffusion Tensor Imaging; functional Magnetic Resonance Imaging; Language Recovery; Left Middle Cerebral Artery Stroke; Nonfluent Aphasia
MeSH Terms: conditions — Aphasia; Aphasia, Broca; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic Stroke patients with Nonfluent Aphasia: patients with left hemisphere (LH) stroke who have chronic nonfluent aphasia

SUMMARY:
The purpose of this research is to utilize functional magnetic resonance imaging (fMRI) to investigate brain reorganization for language behavior in stroke patients with aphasia. A primary focus of the study is on recovery of nonfluent propositional speech and naming in chronic aphasia patients. The fMRI technique is used to examine activation in the left hemisphere (LH) and right hemisphere (RH), during recovery of specific language behaviors in chronic nonfluent aphasia patients.

DETAILED DESCRIPTION:
PURPOSE: The purpose of this 4-year fMRI research is to study brain reorganization for language in patients with left hemisphere (LH) stroke who have chronic nonfluent aphasia. This fMRI research is fundamental and critical to the PI's NIH RO1 grant, Transcranial Magnetic Stimulation (TMS) to Improve Speech in nonfluent aphasia, which was recently renewed for 5 years, 2006-11. There is no overlap in the studies. The NIH grant provides the TMS (real and sham). This VA grant provides 4 different fMRI tasks performed pre- and post- a series of TMS treatments (real and sham) - Overt Naming fMRI; Overt Propositional Speech fMRI; and Nonverbal Semantic Decision tasks for Nouns, and for Actions.

The investigators have observed that application of TMS to an anterior portion of right (R) Broca's homologue (pars triangularis, PTr), results in significantly improved picture naming ability at 2 and 8 Mo. after the last (10th) TMS treatment, in aphasia patients who began TMS at 5-11 years poststroke. Also, half of these nonfluent aphasia patients improved their Phrase Length in propositional speech, post-TMS.

RATIONALE: The investigators and others have observed that patients with chronic, nonfluent aphasia (poor, hesitant speech) have overactivation of R hemisphere (RH) cortical language homologues. The investigators hypothesize this represents a maladaptive plasticity and probably poor active inhibition during speech. Slow, 1 Hz TMS can be used to suppress cortical excitability. The goal is to use 1 Hz TMS to inhibit/suppress the overactivation in RH language homologues. The investigators' early TMS research has shown that suppression of R PTr in these patients is associated with improved speech. The fMRI studies proposed in this VA grant will help to investigate the neurophysiological changes underlying improvement post- TMS in propositional speech and in nonverbal semantic decision tasks. The new MRI technique, diffusion tensor imaging (DTI) will be used to study WM pathways subjacent to cortex treated with TMS.

DESIGN: Randomized, sham-control, incomplete crossover design with 32 patients (16 mild-moderate; 16 severe nonfluent), half receive real TMS series only; half, sham TMS 1st, and real 2nd. Language, Neuropsych. testing, and fMRIs are performed at Entry, and at 2 Mo. post-10 real or sham TMS treatments; and at 6 Mo. post real. There are 4 Projects: 1) fMRI during overt naming and propositional speech (Overt Picture Naming and Picture Descriptions/Story Telling; 2) fMRI during a Nonverbal Semantic Decision Task with Superordinate Noun Icons; 3) fMRI during a Nonverbal Semantic Decision Task with Action and Object Icons; 4) DTI. DTI is performed only at Entry (all subjects). Normal controls (n=8) do not receive TMS; they are studied with fMRI at Entry, at 2 and 6 Mo. later.

HYPOTHESES: Following the real TMS to suppress R PTr, there will be less overactivation on fMRI (better modulation) in RH language homologues, and new LH activation (including L perilesional areas and L SMA). This will be associated with improved propositional speech (BDAE) and nonverbal semantic decision ability at 2 and 6 Mo. post-real TMS. No language or fMRI changes are expected post-sham TMS. The fMRIs performed 3x with the normal controls are not expected to show change, but will document the neural networks for the fMRI tasks.

ELIGIBILITY:
Inclusion Criteria:

* Aphasia patients with a single, unilateral, left hemisphere stroke.
* Patients must be native speakers of English
* Patients must be at least 6 months poststroke and produce mild-severe nonfluent speech. Minimum Language requirements: 2-4 word phrase length on elicited propositional speech
* Auditory Comprehension a the 25th percentile or higher on the BDAE subtests for Word Comprehension and Commands, sufficient to cooperate during testing
* The ability to name a minimum of 3 items on the Boston Naming Test at entry into study.
* Patients must understand the nature of the study and give informed consent.
* Normal right-handed controls with no history of neurological disease or substance abuse; age, education and gender-matched to the Aphasia cases.

Exclusion Criteria:

* Patients with more than one stroke in the left hemisphere or patients with bilateral strokes.
* Each participant must be able to have an MRI scan.
* MRI is contraindicated for pregnant women.
* Patients will be excluded if they have the following:
* Intracranial metallic bodies from prior neurosurgical procedure, implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit or ventriculoperitoneal shunt
* Past history of seizures within one year or unexplained loss of consciousness Family history of epilepsy
* Acute, unstable medical conditions
* History of substance abuse (within last 6 months)
* Abnormal neurological exam, other than as signs of the condition being studied
* Abnormal MRI, or history of known structural brain abnormality other than as signs of the condition studied in the present protocol.
* Administration of investigational drug within 5 halflives of the drug prior to testing.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic stroke patients with nonfluent aphasia
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 1999-10-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Cerebral Activation in the Left and Right Brain Hemispheres | Out to 6 months, from baseline entry
  Cerebral Activation in the Left and Right Brain Hemispheres

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Naeser, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Naeser MA, Martin PI, Baker EH, Hodge SM, Sczerzenie SE, Nicholas M, Palumbo CL, Goodglass H, Wingfield A, Samaraweera R, Harris G, Baird A, Renshaw P, Yurgelun-Todd D. Overt propositional speech in chronic nonfluent aphasia studied with the dynamic susceptibility contrast fMRI method. Neuroimage. 2004 May;22(1):29-41. doi: 10.1016/j.neuroimage.2003.11.016. PMID 15109995
- [Result] Martin PI, Naeser MA, Theoret H, Tormos JM, Nicholas M, Kurland J, Fregni F, Seekins H, Doron K, Pascual-Leone A. Transcranial magnetic stimulation as a complementary treatment for aphasia. Semin Speech Lang. 2004 May;25(2):181-91. doi: 10.1055/s-2004-825654. PMID 15118944
- [Result] Martin PI, Naeser MA, Ho M, Doron KW, Kurland J, Kaplan J, Wang Y, Nicholas M, Baker EH, Alonso M, Fregni F, Pascual-Leone A. Overt naming fMRI pre- and post-TMS: Two nonfluent aphasia patients, with and without improved naming post-TMS. Brain Lang. 2009 Oct;111(1):20-35. doi: 10.1016/j.bandl.2009.07.007. Epub 2009 Aug 19. PMID 19695692
- [Result] Martin PI, Naeser MA, Ho M, Treglia E, Kaplan E, Baker EH, Pascual-Leone A. Research with transcranial magnetic stimulation in the treatment of aphasia. Curr Neurol Neurosci Rep. 2009 Nov;9(6):451-8. doi: 10.1007/s11910-009-0067-9. PMID 19818232
- [Result] Naeser MA, Martin PI, Lundgren K, Klein R, Kaplan J, Treglia E, Ho M, Nicholas M, Alonso M, Pascual-Leone A. Improved language in a chronic nonfluent aphasia patient after treatment with CPAP and TMS. Cogn Behav Neurol. 2010 Mar;23(1):29-38. doi: 10.1097/WNN.0b013e3181bf2d20. PMID 20299861
- [Result] Kaplan E, Naeser MA, Martin PI, Ho M, Wang Y, Baker E, Pascual-Leone A. Horizontal portion of arcuate fasciculus fibers track to pars opercularis, not pars triangularis, in right and left hemispheres: a DTI study. Neuroimage. 2010 Aug 15;52(2):436-44. doi: 10.1016/j.neuroimage.2010.04.247. Epub 2010 May 8. PMID 20438853
- [Result] Naeser MA, Martin PI, Treglia E, Ho M, Kaplan E, Bashir S, Hamilton R, Coslett HB, Pascual-Leone A. Research with rTMS in the treatment of aphasia. Restor Neurol Neurosci. 2010;28(4):511-29. doi: 10.3233/RNN-2010-0559. PMID 20714075
- See also: VA Boston Healthcare System Research Service Website — http://www.boston.va.gov/
- See also: The Harold Goodglass Aphasia Research Center is a service of the National Institute on Deafness and Other Communication Disorders — http://www.bu.edu/aphasia
- See also: Website for The Aphasia Research Lab of Margaret Naeser, Ph.D., VA Boston Healthcare System and Boston University School of Medicine — http://www.bu.edu/naeser/aphasia